CLINICAL TRIAL: NCT05116579
Title: Circulating Tumor DNA (ctDNA) Monitoring in the Assessment and Prediction of the Efficacy of PARP Inhibitors (PARPi)
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonghong Li, Deputy Director of the Department of Urology, Sun Yat-sen University
Other Study IDs: 2021-FXY-171
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Whole blood and tumor tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the application value of customized ctDNA monitoring in efficacy assessment and prediction during PARPi treatment

DETAILED DESCRIPTION:
This clinical study is an open-label, single-center, observational study to evaluate the application value of customized ctDNA monitoring in efficacy assessment and prediction during PARPi treatment in mCRPC patients. A total of 30 participants with second-line treatment failure will be registered in this study. Whole blood collection will be conducted during the treatment for ctDNA detection, homologous recombination repair (HRR) genes testing, personalized panel customization and whole exome sequencing.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the following criteria:

1. Willing and able to provide informed consent.
2. Adult males from 18 to 75 years age.
3. History of histologically or cytologically confirmed adenocarcinoma of the prostate with Homologous Recombination Deficiency or DDR genes mutation (BRCA1/2, ATM, BARD1, BRIP1, CDK12, CHEK1, CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, RAD54L) detected by high throughput sequencing
4. Documented evidence of metastatic castration resistant prostate cancer (mCRPC) and proposed treatment of PARP inhibitors.
5. Evidence of measurable target lesion in imaging studies.
6. Participants can provide adequate formalin fixed paraffin-embedded (FFPE) tumor tissue collected before any treatment: tumor cell content>30% and necrotic cells<10%.
7. ECOG performance status 0-1
8. Estimated survival≥12 weeks

Exclusion Criteria:

Patients must NOT meet any of the following criteria:

1. Do not meet the inclusion criteria.
2. Under any other anti-tumor therapy like chemotherapy and/or immunotherapy.
3. Receiving organ transplantation in the last 3 months.
4. Participants with autoimmune diseases or history of HBV, HCV or HIV infection (acute or chronic).
5. Participants with pneumonia.
6. Severe concurrent illness or co-morbid disease that would make the subject unsuitable for enrolment
7. Unwilling and unable to provide informed consent.
8. Patients who are judged unsuitable for clinical trial participation by the investigators.

Elimination Criteria:

Violation of the prescribed rule of medication that may influence the judgment of curative effect and safety.

Ages: 18 Years to 75 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: clinic-based sample
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-31 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Radiological progression free survival (rPFS) | From date of randomisation to until radiographic progression (up to 1 year)
  Radiological progression free survival (rPFS) - defined as the time from randomisation to radiological progression, assessed by investigator per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 (soft tissue) and Prostate Cancer Working Group-3 (PCWG-3) criteria (bone), or death from any cause, or the last follow-up, whichever occurs first
Objective Response Rate (ORR) | From randomisation until radiographic progression (up to 1 year)
  ORR is the percentage of patients with at least one visit response of Complete response (CR) or Partial response (PR), in their soft tissue disease assessed by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), in the absence of progression on bone scan assessed by Prostate Cancer Working Group 3 (PCWG3)). Per RECIST v1.1, CR=Disappearance of all target lesions; PR = >=30% decrease in the sum of diameters of target lesions; For each treatment group, ORR is the number of patients with a CR and PR.
PSA response rate | From randomisation until radiographic progression (up to 1 year)
  PSA response rate is defined as the proportion of patients with a PSA decline (defined as a ≥30%, ≥50% and other declines in PSA from baseline).

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  OS is defined as time from treatment commencement to death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yonghong Li, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China